CLINICAL TRIAL: NCT04149756
Title: An Observation Study on Maintaining Weight for 6 Months After 3 Months of Weight Loss Program
Brief Title: Persistent Weight Maintenance for 6 Months After 3 Months of Active Weight Loss
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-Won Lee, Professor, Gangnam Severance Hospital
Other Study IDs: YI201905
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Weight Reduction
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood 20ml, serum, plasma, peripheral blood mononuclear cell
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- overweight or obese adults: overweight or obese adults who participate the trial (NCT03675191)
  Interventions: Other: observation of weight after 6months

INTERVENTIONS:
Other: observation of weight after 6months — This study is an observational study for 96 people who have completed the previous weight loss program.
  We will check the body composition and lipid profile of the participants who voluntarily visit after 6months after the end of the study. .

SUMMARY:
This study is intended to report changes in the weight and metabolic indicators of the subjects six months after the end of the study for adults with a risk factor of 27 kg/m2 or higher (formerly the research task name[clinicaltrial.gov;NCT03675191]).

DETAILED DESCRIPTION:
There was no special intervention after the previous research intervention. After the previous research was completed, we will check the changes in the body composition and metabolic indicators over six months.

ELIGIBILITY:
Inclusion Criteria:

* Those who have participated in the previous trial (NCT03675191) and have completed the three-month study
* Those who agreed the trial.

Exclusion Criteria:

* Those who have withdrawn the previous trial (NCT03675191)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Body mass index (BMI) more than 27kg/m2 with comorbidities or BMI more than 30kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
weight | after 6months
  weight changes

SECONDARY OUTCOMES:
lipid profile | after 6months
  total cholesterol, LDL cholesterol, HDL cholesterol, triglyceride

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jin Kwon, Dr, Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance hospital, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No